CLINICAL TRIAL: NCT01467193
Title: The Effect of Dietary Fat Load and Physical Exercise on the Flexibility and Partitioning of Ectopic Lipids.
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Prof. Dr. med E. Christ, MD, PhD, Division of Endocrinology, Diabetes and Clinical Nutrition, Univeristy Hospital Bern
Other Study IDs: 234/10
Record Dates: First submitted 2011-11-03; First posted 2011-11-08 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Ectopic Lipids; Insulin Sensitivity; Aerobic Exercise; Fat Load; Growth Hormone Deficiency
MeSH Terms: conditions — Insulin Resistance; Dwarfism, Pituitary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: Endurance trained athletes: minimal >50 mlO2/KG body weight
- 2: Sedentary healthy control subjects: age, BMI, Gender and waist matched (to the growth hormone deficient patients)
- 3: GHD patients without a GH substitution therapy in the last 6 months
  Interventions: Dietary Supplement: Fat diet; Other: 2h standardized aerobic exercise

INTERVENTIONS:
Dietary Supplement: Fat diet — Instructions for a high fat diet will be given at the end of visit 2. This consists of the usual food intake with a supplementary fat intake of 0.75g fat/kg BW, administered as 3 additional snacks. These snacks will be distributed in pre-packed bags. A food diary will be kept. All arms will receive this diet during the 3 days preceding the clamp.
  Groups: 3
Other: 2h standardized aerobic exercise — Aerobic (50-60% of Vo2 max) standardized exercise on a bicycle during 2 hours
  Groups: 3

SUMMARY:
This study aims at assessing the effect of standardized dietary fat load and short-term aerobic exercise on systemic lipolysis, flexibility and partitioning of ectopic fat stores (intramyocellular = IMCL, intrahepatocellular = IHCL, intramyocardial lipids = IMCaL) in relation to FFA in endurance trained athletes and hypopituitary patients compared to sedentary healthy control subjects.

Exercise is a powerful stimulation for growth hormone (GH) secretion in health. A standardised exercise test can, therefore, be discriminative for the diagnosis of GH-deficiency in adults. This will be assessed.

Hypothesis (ectopic fat stores)

1. Ectopic fats stores are flexible fuel stores and are influenced by diet and physical activity.FFA availability may play an important regulatory role.
2. There is a tissue specific partitioning of triglycerides and/or FFA among non-adipose organs after fat load and physical exercise
3. The flexibility of ectopic fat stores is related to insulin sensitivity
4. Lipolytic and anti-lipolytic hormones are critical for regulating FFA availability (at rest or during exercise) and therefore also for the regulation of ectopic fat stores.
5. GH is a lipolytica hormone. Lack of GH in adulthood is related to decreased FFA availability thereby influencing ectopic lipid stores Hypothesis diagnosis of GHD
6. A short intensive physical exercise shows a good discriminative power to diagnose GHD.

DETAILED DESCRIPTION:
Background

Obesity, in particular visceral obesity, is associated with impaired insulin action on target tissues (insulin resistance or metabolic syndrome) that, in turn, is related to an increased risk for cardiovascular mortality and morbidity. Pathophysiological mechanism remains unclear. Interventions in patients with impaired glucose tolerance/impaired fasting glucose have consistently demonstrated that by increasing physical activity and reducing calorie intake the risk to convert to frank type 2 diabetes is decreased, even more efficiently than by early medical therapy with metformin.

Physically inactive and overweight subjects do not only store the excess of fat in the intra-abdominal or subcutaneous department but also in non-adipose tissue (="ectopic" tissues), such also skeletal muscle, liver and myocardium, also called intramyocellular lipids (IMCL), intrahepatocellular lipids (IHCL) and intramyocardial lipids (IMCaL).This ectopic lipid accumulation occurs either by increased free fatty acids (FFA) uptake, increase synthesis in the involved tissues or reduced FFA oxidation.

The relative contribution of these factors to ectopic lipid accumulation varies in different physiological conditions (i.e. physical exercise, fasting, postprandial condition) and in different tissues. In addition, it may be influenced by hormones that regulate lipid metabolism. There is increasing evidence that ectopic fat and its intermediate metabolites interfere with insulin signalling, thereby contributing to the impaired insulin action on target tissues such as liver and skeletal muscle. It has been well showed that high fat oxydation capacity allows to keep a lower lipolytic activity and therefore low levels of lipolyse degradation products. Strong evidence is accumulating that these intermediates interact with insulin signalling finally resulting in insulin resistance.

There is still scarce data about the behaviour of ectopic fat stores in the presence of positive(nutritional fat excess) or negative energy balance (physical activity) and the role of hormones in regulating these fat depots.

Additionally,we have previously shown that GH values obtained during a 2h standardized aerobic exercise of moderate intensity revealed a high diagnostic accuracy in predicting severe GHD in adult individuals. Whether a shorter exercise on higher intensity may lead to comparable results has to be assessed.

Objective

The study aims to comprehensively assess the flexibility and partitioning of ectopic fat deposition and to define the role of relevant hormones (especially GH and insulin) in relation to the availability of FFAs as well as their role in the process of ectopic fat deposition and consumption. Another objective is to investigate the role of a standardized fat load and aerobic exercise on IMCaL.

Methods

Using the two-step hyperinsulinaemic-euglycaemic clamp technique hepatic and peripheral insulin sensitivity is assessed.

Lipid depots (skeletal muscle and liver) are repeatedly measured by MR-spectroscopy, subcutaneous and visceral fat mass by whole body MR-imaging.

Exercise capacity ist measured on a bicycle (incl. spiroergometry). Counterregulatory hormones, glucose and free fatty acids are measured during a 2h physical exercise at 50-60 VO2max.

Blood samples to evaluate GH will be taken immediately before and after the Vo2 max-test, as well as 15, 30 and 45minutes after the end of the exercise test.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients >18 years old
* Capable to exercise for 120 minutes on a treadmill
* Willingness to participate in the study and to give written consent.
* Normal ECG during ergometry
* Specific for Athletes: VO2max> 50 ml/kg/min
* Specific for GHD patients: no GH substitution in the last 6 months
* Specific for sedentary controls: Matched the GHD patients for age, gender, BMI and waist

Exclusion Criteria

* Abnormal liver or renal function
* Active neoplasia
* Severe cardiovascular disease (unstable coronary artery disease, heart failure NYHA III-IV)
* Haemophilia
* Inability to exercise
* Contraindications to exposure to a 3 T magnetic field
* Abnormal ECG during ergometry
* Women in childbearing age unless on a continuous contraceptive therapy or surgically sterilized
* Depression, psychosis and other severe personality disorders
* Pregnant women
* Excessive alcohol consumption (>60g/d) or drug abuse

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Athletes:Endurance trained athletes: minimal >50 mlO2/KG body weight
  GH-deficient adult patients: NO GH-replacement therapy during the last 6 months
  Sedentary controls: age, BMI, Gender and waist matched (to the growth hormone deficient patients) healthy control subjects
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2011-08; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Flexibility of IMCaL, IMCL and IHCL (fat load and exercise) | Year 1 to 4

SECONDARY OUTCOMES:
Determination of visceral fat mass by MRI | Year 1 to 4
Determination of peripheral and hepatic insulin sensitivity by two step hyperinsulinemic euglycemic clamp | Year 1 to 3
maximal exercise capacity | Year 1 to 3

CONTACTS AND LOCATIONS:
Overall Officials: Emanuel Christ, Prof. Dr med. MD, PhD, Principal Investigator — Division of Endocrinology, Diabetes and Clinical Nutrition, University Hospital Bern
Locations (1):
- Department of Endocrinology, Diabetes and Clinical Nutrition, University Hospital Bern, Bern, Switzerland

REFERENCES:
- [Result] Zueger T, Alleman S, Christ ER, Stettler C. Exercise-induced GH secretion in the assessment of GH deficiency in adult individuals. Eur J Endocrinol. 2011 Nov;165(5):723-8. doi: 10.1530/EJE-11-0539. Epub 2011 Aug 19. PMID 21856788
- [Derived] Loher H, Jenni S, Bucher J, Krusi M, Kreis R, Boesch C, Christ E. Impaired repletion of intramyocellular lipids in patients with growth hormone deficiency after a bout of aerobic exercise. Growth Horm IGF Res. 2018 Oct-Dec;42-43:32-39. doi: 10.1016/j.ghir.2018.08.001. Epub 2018 Aug 17. PMID 30153529